CLINICAL TRIAL: NCT06386419
Title: A Real-world, Prospective, Multi-center, Open-label, Phase 4 Clinical Study to Evaluate the Safety and Effectiveness of Subcutaneous Injection of Inclisiran Sodium in Indian Patients With Primary Hypercholesterolemia or Mixed Dyslipidemia
Brief Title: A Clinical Study to Evaluate the Safety and Effectiveness of Inclisiran Sodium in Indian Patients With Primary Hypercholesterolemia or Mixed Dyslipidemia
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CKJX839A1IN03
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Primary Hypercholesterolemia; Mixed Dyslipidemia
Keywords: Inclisiran,; primary hypercholesterolemia; mixed dyslipidemia; ASCVD; PCSK9; Phase 4
MeSH Terms: interventions — ALN-PCS

STUDY DESIGN:
Intervention Model Description: open label assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- inclisiran (Experimental): 300 mg inclisiran sodium equivalent to 284 mg inclisiran administered as a single SC injection
  Interventions: Drug: inclisiran

INTERVENTIONS:
Drug: inclisiran — Inclisiran sodium 300 mg SC. Three single doses of inclisiran sodium will be administered to the participants on Day 1, Day 90, and Day 270, respectively
  Other Names: KJX839

SUMMARY:
This study is to generate post-marketing safety and effectiveness data of inclisiran sodium in Indian patients as per approved indication i.e., primary hypercholesterolemia (heterozygous familial and non-familial) or mixed dyslipidemia that more closely resembles the real-world population intended to be treated with inclisiran sodium.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm, open-label, interventional Phase 4 clinical study and will be conducted across several sites in India.

The study consists of:

* Open-label treatment period: The open-label treatment period will be of 270 days during which 3 single doses of inclisiran sodium will be administered subcutaneously (SC) on Day 1, Day 90, and Day 270, respectively. On Day 1/Dose 1 visit, the patients will be assessed by the Investigator for their eligibility to receive inclisiran sodium based on their medical history and previous lipid test reports. The study treatment i.e., inclisiran sodium will be prescribed as per the latest India Prescribing Information (PI). The assignment of the participant to the therapy will be decided within the current practice and the medical indication and will clearly be separated from the decision to include the participant in the study.
* Safety follow-up period: The safety follow-up will be performed 30 days after each dose administration of the study treatment i.e., Day 30, Day 120, and Day 300. The follow-up on Day 30 and Day 120 visits will be conducted telephonically while Day 300 visit will be an onsite follow-up visit.

This study will be conducted in compliance with Good Clinical Practices (GCP) including the Declaration of Helsinki and New Drugs and Clinical Trials (NDCT) Rules, 2019 requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female Indian participants aged ≥18 years or older.
2. Participants for whom the treating physician prescribes treatment with inclisiran sodium in adherence with the India PI i.e., patients who are diagnosed with primary hypercholesterolemia (heterozygous familial and non-familial) or mixed dyslipidemia, as an adjunct to diet:

   1. in combination with a statin or statin with other LLTs in patients unable to reach LDL-C goals with the maximum tolerated dose of a statin, or
   2. alone or in combination with other LLTs in patients who are intolerant to statins or for whom a statin is contraindicated.
3. Participants on LLTs should be on a stable dose for ≥30 days before the first dose administration of the study treatment.

Exclusion Criteria:

1. Any surgical and/or medical condition, which in the opinion of the treating physician, may place the participant at higher risk of his/her participation in the study, or is likely to prevent the participant from complying with the requirements of the study or completing the study.
2. Participants who have previous exposure to inclisiran sodium.
3. Pregnant or nursing (lactating) women.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Incidence and type of treatment-emergent adverse events (TEAEs) | 10 months (300 days)
  An Adverse Event (AE) is any untoward medical occurrence in a participant that does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product. A TEAE will be defined as an AE that begins or that worsens in severity after at least 1 dose of the study treatment has been administered.

SECONDARY OUTCOMES:
Mean change in LDL-C from baseline to Day 300. | Baseline, Day 300
  Mean change in LDL-C from baseline to Day 300 to valuate the effectiveness of inclisiran sodium in terms of change in low-density lipoprotein cholesterol (LDL-C) levels.
Proportion of the participants with ≥50% LDL-C reduction on Day 300 | Baseline, Day 300
  Proportion of the participants with ≥50% LDL-C reduction on Day 300 to evaluate the effectiveness of inclisiran sodium in terms of change in low-density lipoprotein cholesterol (LDL-C) levels
Proportion of the participants who attain global lipid targets for their level of atherosclerotic cardiovascular disorders (ASCVD) risk | Day 300
  global lipid targets for their level of ASCVD risk: 55 mg/dL for ASCVD very high-risk participants 70 mg/dL for ASCVD high-risk participants
Percentage change in TC, HDL-C, non-HDL-C, VLDL-C and TG | Baseline, Day 300
  Percentage change in total cholesterol (TC), high-density lipoprotein cholesterol (HDL-C), non-HDL-C, very low-density lipoprotein cholesterol (VLDL-C), and triglycerides (TG) to evaluate the effectiveness of inclisiran sodium in reducing other lipid markers from baseline to Day 300.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- India (7):
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Madurai, Tamil Nadu
  - Novartis Investigative Site, Vellore, Tamil Nadu
  - Novartis Investigative Site, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com